CLINICAL TRIAL: NCT03296150
Title: ADOPT-PRESTAGE: Randomized Controlled Trial on Acceptability, Diffusion and Impact on Treatment Adherence and Persistence of the PRESTAGE Program (Program for Education and Support for Oral Cancer Treatments in the Elderly) - Randomized Controlled Study Evaluating the Impact of the Program PRESTAGE
Brief Title: ADOPT-PRESTAGE: Study Evaluating the Impact of the Program PRESTAGE
Acronym: ADOPT-PRESTAGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL16_0149
Record Dates: First submitted 2017-09-23; First posted 2017-09-28 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Cancer; Oral Anticancer Drugs
Keywords: therapeutic educational program; adherence; quality of life; elderly; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm : Information (No Intervention): Patients will receive the usual standard information delivered to patients
- Intervention arm : Therapeutic educational program (Experimental): Patients will receive the therapeutic educational program "PRESTAGE"
  Interventions: Behavioral: PRESTAGE

INTERVENTIONS:
Behavioral: PRESTAGE — PRESTAGE educational program targets the acquisition by the patients and their caregivers of competencies in (1) a better understanding of their disease and (2) their treatment, (3) a better drug management, including both anticancer and supportive treatments, (4) maintenance of a good nutritional status, (5) general health and psychological well being and (6) physical well being. After an individual educational diagnosis, each patient will be proposed an individualized educational program consisting in 1 to 6 of these workshops. An individualized final interview - entitled educational synthesis - will assess patient's skills and satisfaction.
  Arms: Intervention arm : Therapeutic educational program

SUMMARY:
As the proportion of oral anticancer treatments is continuously increasing, adherence appears as a major issue for patients' outcomes. Poor adherence affects particularly geriatric patients due among others to polypharmacy or cognitive impairment. Thus, the need for educational programs in this population has been regularly emphasized.

PRESTAGE educational program was built after an external and internal analysis of educational needs in elderly patients treated with oral cancer treatments. It implicates a multidisciplinary educational team (nurses, physicians, pharmacists, psychologists, physiologists, social workers...). Six educational workshops were designed with the following endpoints: disease and treatment understanding, treatment management, nutrition and psychological as well as physical well being.

ADOPT-PRESTAGE is a clinical, prospective, interventional, open-label, multicenter, randomized, controlled trial designed to evaluate the impact of PRESTAGE program. It is, to the investigators' knowledge, the first randomized controlled trial evaluating the acceptability and impact (adherence, clinical benefit) of an educational program in an elderly cancer population. The primary endpoint of this trial will be to evaluate adherence using an indirect objective adherence measure: the Medication Event Monitoring System (MEMS). Secondary endpoints include quality of life and evaluation of changes in patients' behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 70 years,
* For which oral anticancer therapy has been initiated within the previous 45 days or will be started within 45 days
* For any type of cancer, solid or hematologic, any stage
* Estimated life expectancy> 6 months
* Affiliation to social security or equivalent
* Patients who can answer questionnaires and protocol evaluations
* Informed consent signed by patients
* Domiciled within 50 km around the investigating center

Exclusion Criteria:

* For patients with breast cancer, exclusive treatment with hormone therapy
* First-generation Hormone Therapy in Prostate Cancer
* Patient not available for regular follow-up whatever the cause (geographic, family, social, psychological)
* Any serious condition, ie serious physical or mental, leading to a disability permanent and likely to prevent the proper course of treatment
* Patient deprived of liberty or under guardianship

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2018-03-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Adherence evaluated by MicroElectronic Monitoring System | at 4 months (after intervention or information)
  Adherence will be evaluated with MicroElectronic Monitoring System. A composite score such as described by Thivat et al. in 2013 will be used.

SECONDARY OUTCOMES:
Adherence evaluated by Morisky questionnaires | 4 months to 12 months
  Results to Morisky questionnaires will be evaluated such as adherence with MEMS, until 12 months.
Adherence evaluated by pharmacy medication refill -based adherence | 4 months to 12 months
  Results to pharmacy medication refill -based adherence will be evaluated such as adherence with MEMS, until 12 months.
Health-related quality of life evaluated by QLQ-C30 quality of life questionnaire | 4 months to 12 months
Health-related quality of life evaluated by the QLQ-ELD14 quality of life questionnaire | 4 months to 12 months
Health-related quality of life evaluated by the EORTC quality of life questionnaire | 4 months to 12 months
Changes in patients' behaviors evaluated by questionnaires | 4 months to 12 months
  Beliefs about Medication questionnaire and satisfaction with medication questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Olivia LE SAUX, Study Chair — Hospices Civils de Lyon
Locations (9):
- France (9):
  - Service de neuro-oncologie, Hôpital Pierre Wertheimer, HCL, Bron
  - Service de Gériatrie, Centre Hospitalier de Givors, Givors
  - Service d'oncologie médicale, Centre Hospitalier Universitaire de Grenbole, La Tronche
  - Service de Médecine du vieillissement, Hôpital Edouard Herriot, HCL, Lyon
  - Service de médecine du vieillissement, Hôpital de la Croix-Rousse, HCL, Lyon
  - Service d'oncologie médicale, Cnetre Léon Bérard, Lyon
  - Service d'oncologie, Centre Hospitalier Annecy Genevois, Metz-Tessy
  - Service de Médecine du vieillissement, Centre Hospitalier Lyon Sud (Hospices Civils de Lyon), Pierre-Bénite
  - service de gériatrie, Hôpital de la Charité, Centre Hospitalier Universitaire de St-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No